CLINICAL TRIAL: NCT02403999
Title: A Clinical Study in Infants to Assess the Tolerability of Three Wash Products
Brief Title: A Tolerability Assessment Study of Three Wash Products in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 203080; RH02709 (Other: GSK)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2017-11

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test shampoo (Experimental): Participants' will be instructed to use the test product as per the label instructions for a minimum of twice per week for 2 weeks.
  Interventions: Other: Test shampoo
- Test bath foam (Experimental): Participants' will be instructed to use the test product as per the label instructions for a minimum of twice per week for 2 weeks.
  Interventions: Other: Test bath foam
- Test head to toe Wash (Experimental): Participants' will be instructed to use the test product as per the label instructions for a minimum of twice per week for 2 weeks.
  Interventions: Other: Test head to toe wash

INTERVENTIONS:
Other: Test shampoo — Participants used Oilatum Soothe & Protect Shampoo at home in place of their usual wash product at least twice weekly for a two week period.
  Arms: Test shampoo
Other: Test bath foam — Participants used Oilatum Soothe & Protect Bath Foam at home in place of their usual wash product at least twice weekly for a two week period.
  Arms: Test bath foam
Other: Test head to toe wash — Participants used Oilatum Soothe & Protect Head to Toe Wash at home in place of their usual wash product at least twice weekly for a two week period.
  Arms: Test head to toe Wash

SUMMARY:
This will be a single centre, evaluator blind, randomized, parallel group, stratified, two week study in healthy participants. The clinical study is designed to provide reassurance that the formulations developed for children and babies with mild to moderately dry skin and for children whose skin is prone to atopic dermatitis (eczema) are well tolerated in the target population, babies and young children with dry skin.

ELIGIBILITY:
Inclusion Criteria:

* Participants up to 18 months of age at the screening/baseline visit with good general health and no major physical disabilities
* Parent/legal guardian reported dry skin
* Voluntary written informed consent form by parent/legal guardian as an evidence to understanding of the study and willingness to participate

Exclusion Criteria:

* Allergy/intolerance or hypersensitivity to the study material or any of their stated ingredients
* Participant with skin condition that warrants medical intervention, current episode of eczema/atopic dermatitis or has had an episode in the 3 months prior to screening, not regular use of moisturizers (variable application frequency)
* Use of oral corticosteroids/immunosuppressive medication within 4 weeks or topical corticosteroids/topical anti-itch products within 2 weeks of baseline
* Child in Care; participants' previous participation in this study/another clinical study/receipt of investigational drug within 30 days of the screening visit
* Parent/legal guardian aged 18 years or under, employee of the sponsor or the study site or members of their immediate family
* Participant living in the same household of an already enrolled participant

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Edinburgh, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were recruited from one center in United Kingdom.
Pre-assignment Details: A total of 32 participants were screened and enrolled in the study, out of which 31 participants were randomized to the study and 1 participant was screening failure as participant did not meet study criteria.
Groups:
- Test Shampoo; Test Bath Foam; Test Head to Toe Wash: Participants were instructed to use the test product as per the label instructions for a minimum of twice per week for 2 weeks.
Period: Overall Study
Arm/Group | Test Shampoo | Test Bath Foam | Test Head to Toe Wash
Started | 10 | 10 | 11
Completed | 10 | 10 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Shampoo | Test Bath Foam | Test Head to Toe Wash | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: Months] | 9.0 (5.62) | 10.9 (4.20) | 10.1 (3.86) | 10.0 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 4 | 16
  Male | 2 | 6 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 10 | 11 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Assessment of Test Products
Description: The tolerability of the test products under normal conditions of use was assessed by the paediatrician using a 5 point scale: where score 1= very good; 2= good; 3= acceptable; 4= poor and 5= very poor.
Time Frame: At Day 14
Population: Safety population (overall): included all the participants who received at least one of the test product. Participants were further divided in two age strata Age <12 months and Age ≥ 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Shampoo | Test Bath Foam | Test Head to Toe Wash
Number analyzed (Participants) | 10 | 10 | 11
Participants
  Overall: Score 1 (Very good) | 9 | 10 | 11
  Overall: Score 2 (Good) | 1 | 0 | 0
  Overall: Score 3 (Acceptable) | 0 | 0 | 0
  Overall: Score 4 (Poor) | 0 | 0 | 0
  Overall: Score 5 (Very poor) | 0 | 0 | 0
  Overall: >3 (Not acceptable) | 0 | 0 | 0
  Age stratum <12 months: number analyzed (Participants) | 5 | 5 | 6
  Age stratum <12 months: Score 1 (Very good) | 5 | 5 | 6
  Age stratum <12 months: Score 2 (Good) | 0 | 0 | 0
  Age stratum <12 months: Score 3 (Acceptable) | 0 | 0 | 0
  Age stratum <12 months: Score 4 (Poor) | 0 | 0 | 0
  Age stratum <12 months: Score 5 (Very poor) | 0 | 0 | 0
  Age stratum <12 months: >3 (Not acceptable) | 0 | 0 | 0
  Age stratum ≥12 months: number analyzed (Participants) | 5 | 5 | 5
  Age stratum ≥12 months: Score 1 (Very good) | 4 | 5 | 5
  Age stratum ≥12 months: Score 2 (Good) | 1 | 0 | 0
  Age stratum ≥12 months: Score 3 (Acceptable) | 0 | 0 | 0
  Age stratum ≥12 months: Score 4 (Poor) | 0 | 0 | 0
  Age stratum ≥12 months: Score 5 (Very poor) | 0 | 0 | 0
  Age stratum ≥12 months: >3 (Not acceptable) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Overall Dry Skin [ODS] Score at Day 14 (Visual Assessment of Skin)
Description: The changes in participants' skin condition was assessed using the ODS score: where 0= Absent; 1= Faint scaling, faint roughness and dull appearance; 2= Small scales in combination with a few larger scales, slight roughness, whitish appearance; 3= Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks; 4= Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks.
Time Frame: At baseline and day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Shampoo | Test Bath Foam | Test Head to Toe Wash
Number analyzed (Participants) | 10 | 10 | 11
Score on scale
  Overall | -1.2 (0.79) | -0.9 (0.57) | -0.5 (0.69)
  Age Stratum <12 months: number analyzed (Participants) | 5 | 5 | 6
  Age Stratum <12 months | -0.8 (0.84) | -1.0 (0.71) | -0.7 (0.52)
  Age Stratum ≥12 months: number analyzed (Participants) | 5 | 5 | 5
  Age Stratum ≥12 months | -1.6 (0.55) | -0.8 (0.45) | -0.4 (0.89)

ADVERSE EVENTS:
Time Frame: Up to 14 days (± 2 days)
Arm/Group | Test Shampoo | Test Bath Foam | Test Head to Toe Wash
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Shampoo (N=10) | Test Bath Foam (N=10) | Test Head to Toe Wash (N=11)
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.